CLINICAL TRIAL: NCT04434846
Title: Investigating the Sylvatic Transmission and Reservoir Potential of Zika, Dengue, and Chikungunya Viruses of Co-located Humans and Long-tailed Macaques of Thailand and Cambodia
Brief Title: Sylvatic Transmission of Zika, Dengue, and Chikungunya Viruses in Thailand and Cambodia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920054; 20-I-N054
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2021-05-07

CONDITIONS: Dengue Fever; Zika; Vector-Borne Diseases; Chikungunya
Keywords: Vector-Borne Diseases; Arbovirus; Serological Survey; Seroprevalence; Southeast Asia; Natural History
MeSH Terms: conditions — Dengue; Zika Virus Infection; Vector Borne Diseases; Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sera from macaques and humans

GROUPS / COHORTS (1):
- 1: Healthy Cambodian Adults aged 18-55 were screened for antibodies to ZIKV, DENV, and CHIKV at a single time point at Amphae Phnom, Chbar Mon, Cambodia.

SUMMARY:
Background:

Zika, dengue, and chikungunya are spread by mosquitos. These diseases have a major impact on public health. This is especially true in in Southeast Asia. Non-human primates (such as macaques) could play an essential role in spreading these diseases. Researchers want to further understand the relationship between humans and these primates. They want to see how this affects how mosquito-borne viruses are spread in Southeast Asia.

Objective:

To describe the prevalence of Zika virus, dengue virus, and chikungunya virus in the blood of people who live close to long-tailed macaques in Thailand and Cambodia.

Eligibility:

Healthy people aged 18-55 who have lived or worked within approximately 10 kilometers of the Wat Amphae Phnom monkey habitat in Kampong Speu, Cambodia, for a minimum of 2 years

Design:

Participation will last 1 day.

Participants will be screened in person through an interview. Their medical history will be reviewed.

Participants will give information about themselves. This will include sex, age, and behaviors related to the spread of mosquito-borne disease. For example, they will be asked about the number of water containers at their home. They will be asked about recent travel. They will be asked about the extent of their contact with the macaques.

Participants will give a blood sample....

DETAILED DESCRIPTION:
Arboviral epidemics continue to emerge suddenly and spread of disease is unpredictable. The 2015-16 Zika epidemic resulted in a high case number in Thailand, but not in neighboring Cambodia. It is known that nonhuman primates (NHPs) are important reservoirs of arboviruses, but the importance of their epidemiological role in the transmission of arboviruses is not clearly understood. While transmission dynamics are complex and require consideration of many variables, primate reservoirs are not routinely sampled, particularly in Southeast Asia, because of the level of operational complexity and skill required.

Here, we propose a serological survey for evidence of Zika virus (ZIKV), dengue virus (DENV), and chikungunya virus (CHIKV) exposure in long-tailed macaques and human adults who live or work in close proximity to these monkeys in Thailand and Cambodia. We hypothesize that ZIKV seroprevalence in both humans and macaques will be higher in Thailand than Cambodia. With the current rise of arboviral diseases around the world, we hope the results of this study contribute to better understanding of the epidemiology and burden of arboviral diseases in this region.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated ICF
2. Able to provide informed consent
3. Stated willingness to comply with study procedures
4. Male or female, aged 18-55 years
5. Live/work within approximately 10 km of the Wat Amphae Phnom monkey habitat for minimum of 2 years
6. In good general health as evidenced by screening medical history
7. Willing to allow biological samples to be stored for future research

EXCLUSION CRITERIA:

1. Any underlying, chronic, or current medical condition that, in the opinion of the investigator, would interfere with participation in the study (e.g., inability or great difficulty in drawing blood)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy male or female volunteers from Chbar Mon, Cambodia who live or work within approximately 10 km of long-tailed macaque habitats for a minimum of 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Yek, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Malaria Center, Phnom Penh, Cambodia

REFERENCES:
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Ruchusatsawat K, Wongjaroen P, Posanacharoen A, Rodriguez-Barraquer I, Sangkitporn S, Cummings DAT, Salje H. Long-term circulation of Zika virus in Thailand: an observational study. Lancet Infect Dis. 2019 Apr;19(4):439-446. doi: 10.1016/S1473-3099(18)30718-7. Epub 2019 Feb 27. PMID 30826189
- [Background] Weaver SC, Lecuit M. Chikungunya virus and the global spread of a mosquito-borne disease. N Engl J Med. 2015 Mar 26;372(13):1231-9. doi: 10.1056/NEJMra1406035. No abstract available. PMID 25806915

RESULTS

PARTICIPANT FLOW:
Groups:
- Cambodian Adults in Observational Cross-Sectional Study of Arboviral Exposure: Healthy Cambodian Adults of ages 18-55 screening for exposure to ZIKV, DENV, and/or CHIKV. To clarify, no THAI adults were enrolled under this protocol.
Period: Overall Study
Arm/Group | Cambodian Adults in Observational Cross-Sectional Study of Arboviral Exposure
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cross Sectional Enrollment of 300 Adults: Adults of ages 18-55 with ZIKV, DENV, and/or CHIKV seroprevalence living near Amphae Phnom, Cambodia
Arm/Group | Cross Sectional Enrollment of 300 Adults
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 300
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 300
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Cambodia | 300

OUTCOME MEASURES:

1. Primary Outcome: Assessment of DENV, ZIKV, CHIKV Seroprevalence Via Screening PRNT50 Titers in Cambodian Adults.
Description: Proportion of Participants with DENV, ZIKV, CHIKV Seroprevalence Via Screening PRNT50. Outcome will be analyzed unadjusted and adjusted for age, location, vector exposure, and sylvatic reservoir exposure.
Time Frame: 300 at day 0
Measure: Count of Participants; unit: Participants
Groups:
- Cross Sectional Enrollment of 300 Adults: Adults of ages 18-55 with ZIKV antibodies living near Amphae Phnom, Cambodia
Arm/Group | Cross Sectional Enrollment of 300 Adults
Number analyzed (Participants) | 300
Participants | 300

2. Secondary Outcome: Comparative Assessment of Seroprevalence Via PRNT50 Titers for ZIKV, DENV, and CHIKV in Cambodian Adults to That of Thai Adults.
Description: Understanding how the prevalence of these Aedes transmitted viruses differs across the Mekong region is critical for cross-border disease detection and management, particularly given the high level of human migration in the Greater Mekong Subregion.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Cambodian Human Adults: Healthy Cambodian Adults aged 18-55 at a single time point at Amphae Phnom, Chbar Mon, Cambodia.
Arm/Group | Cambodian Human Adults
Number analyzed (Participants) | 300
Participants | 300

3. Secondary Outcome: Assessment of Reactivity to Salivary Gland Homogenate of Aedes Aegypti as Detected by ELISA or Western Blot in Human Sera.
Description: Characterizing vector salivary protein reactivity profiles (mosquitos, ticks, fleas) in Cambodians with vector- borne disease is the first step to better understanding transmission patterns, responsible vectors, and Cambodians' risk of exposure to these vectors.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Cambodian Human Adults
Number analyzed (Participants) | 300
Participants | 300

ADVERSE EVENTS:
Time Frame: This was a cross sectional bioprocurement protocol with a one-time blood draw. Adverse events were monitored on that day, participants exited the study the same day but were always able to call study team - up to three months after study exit - should an adverse event have occurred from a low-risk procedure such as phlebotomy. The enrollment and monitoring period was during the month of February 2020.
Groups:
- 300 Adults Ages 18-55 With ZIKV, DENV, and/or CHIKV Seroprevalence.: Adults ages 18-55 with ZIKV, DENV, and/or CHIKV seroprevalence.
Arm/Group | 300 Adults Ages 18-55 With ZIKV, DENV, and/or CHIKV Seroprevalence.
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04434846/Prot_SAP_ICF_000.pdf